CLINICAL TRIAL: NCT07260786
Title: A Study on the Correlation Between Visual Quality After SMILE and LASEK Procedures and the Visual Conduction Pathways in Patients With Moderate to Low Myopia
Brief Title: the Correlation Between Visual Quality After SMILE and LASEK in Patients With Moderate to Low Myopia
Acronym: SMILE LASEK
Status: Completed | Type: Observational
Sponsor: yuhao shao (Other)
Responsible Party: Sponsor-Investigator, yuhao shao, DR, Tongji University
Organization: Tongji University (Other)
Other Study IDs: 20251022VEP; YNCR2C004 (Other Grant/Funding Number: Tongji University)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Myopia
Keywords: myopia; SMILE; LASEK; VEP; CS
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SMILE: undergoing SMILE
- LASEK: undergoing SMILE

SUMMARY:
1. Study the changes in subjective visual quality, contrast sensitivity, and total ocular aberrations of patients with low-to-moderate myopia after SMILE and LASEK surgeries at different age groups;
2. Evaluate the effects of SMILE and LASEK surgeries on the visual conduction pathway PVEP in patients with refractive errors of different age groups;
3. Clarify the correlations between subjective and objective visual quality after SMILE and LASEK surgeries in patients with refractive errors of different age groups and PVEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractive errors who were scheduled to undergo SMILE surgery and LASEK surgery were selected. The preoperative equivalent spherical diopter (SE) of the affected eye was less than -6D. The surgical plan was based on voluntary principle and was divided into the SMILE group and the LASEK group. Each surgical group was further divided according to age into groups of ≤ 20 years old, 21-30 years old, 31-40 years old, and ≥ 41 years old. Each group consisted of 35 patients. There were no significant differences in gender, equivalent spherical diopter (SE), optical zone, and preoperative best corrected visual acuity among the groups.

Exclusion Criteria:

* The nearsightedness has increased by more than 1D in the past two years. Severe dry eye syndrome, keratoconus, glaucoma, history of eye surgery, severe systemic connective tissue or autoimmune diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People with mild to moderate myopia who have undergone SMILE or LASEK surgeries
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity | Before the operation, 1 week after the operation, 1 month after the operation, 3 months after the operation, 6 months after the operation
  Under sufficient correction conditions, dark adaptation lasted for 10 minutes. Using the CSV-1000 contrast sensitivity tester at a distance of 3 meters, under the conditions of bright vision (85 cd/m ²), bright glare (135 lx), dark vision (3 cd/m ²), and dark glare (28 lx) respectively, Test the highest CS level that can be distinguished at 3, 6, 12 and 18 c/d spatial frequencies one by one. At each spatial frequency, the examinee needs to point out the bar grid sight in the upper and lower two circular sight targets and report the direction of the bar grid. After the result is correct, gradually reduce the bar grid contrast until the examinee can no longer recognize it. The inverse of the lowest recognizable contrast at this time is the contrast sensitivity. Record in logarithmic units according to the grade value conversion table.
VEP | Before the operation, 1 week after the operation, 1 month after the operation, 3 months after the operation, 6 months after the operation
  The VEP examination was repeated forN75 and P100. N75 latency and P100 amplitude and latency scores were calculated on the average waveform. It required manual definition of the lowest negative peak (N75) before P100 peak.
  Amplitude was scored as the difference between these two points and latency was scored as the time difference between N75 lowest peak or P100 peak and stimulus onset.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No